CLINICAL TRIAL: NCT02396836
Title: Randomised Controlled Trial of the Effectiveness of Two Hand Hygiene Techniques Using Alcohol Based Hand Rub on Hand Surface Coverage and Reducing Bacterial Hand Contamination
Brief Title: Randomised Controlled Trial (RCT) of 6 Versus 3 Steps for Hand Hygiene
Acronym: SHoRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: University of Strathclyde (Other); University of East Anglia (Other); NHS Greater Glasgow and Clyde (Other); Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Jacqui Reilly, Professor Jacqui Reilly, Glasgow Caledonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12-170; SIRN04 (Other Grant/Funding Number: Scottish Infection Research Network)
Record Dates: First submitted 2014-08-15; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Hand Hygiene
Keywords: Hand hygiene; Hand decontamination; Microbial load; Hand coverage; Glove juice technique; Ayliffe technique; 6 step technique
MeSH Terms: interventions — Hand Hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 step hand hygiene technique (Active Comparator): Hand decontamination with alcohol hand rub using the World Health Organisations 6 step technique
  Interventions: Other: 6 step technique
- 3 step hand hygiene technique (Experimental): Hand decontamination with alcohol hand rub using the 3 step technique
  Interventions: Other: 3 step technique

INTERVENTIONS:
Other: 6 step technique — Hand decontamination with alcohol hand rub using the World Health Organizations 6 step technique
  Other Names: World Health Organisation 6 step technique for hand hygiene
  Arms: 6 step hand hygiene technique
Other: 3 step technique — Hand decontamination with alcohol hand rub using the 3 step technique
  Other Names: 3 step technique for hand hygiene
  Arms: 3 step hand hygiene technique

SUMMARY:
The aim is to compare the effectiveness of the 6 step hand rub technique versus 3 step hand rub technique in hand coverage and in reducing bacterial contamination on the hands of healthcare workers in practice.

Research questions

1. What is the effectiveness of the 6 step technique in hand coverage compared to the 3 step technique?

   1. What are the most frequently missed sites in hand surface coverage using 6 steps compared to 3 steps?
   2. What is the reduction in bacterial contamination of the hand with the 6 step compared to the 3 step technique?
2. Does site missed or coverage relate to bacterial load?
3. What is the time taken for 6 step technique versus 3 step technique?

DETAILED DESCRIPTION:
The 6 step for decontamination of healthcare workers hand is recommended by the World Health Organization but the 3 step technique is easy to perform and has been shown by some studies to be effective. Compliance with the 6 step technique is not optimum. If the 3 step was more as or more effective than the 6 step compliance with it could be compared with that for the 6 step. No randomised controlled trial comparing the effectiveness of these two techniques using alcohol based hand rub has been conducted.

ELIGIBILITY:
Inclusion Criteria:

* Medical and nursing staff performing a clinical procedure

Exclusion Criteria:

* A procedure requiring use of gloves
* A self declared active skin condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Microbial load on dominant hand | up to 5 min
  A glove juice technique will be used to assess the microbial load on the dominant hand of healthcare workers following use of alcohol hand rub after a clinical procedure.

SECONDARY OUTCOMES:
Hand coverage | up to 5 min
  Ultra violet box will be used to assess hand coverage of the hands of healthcare workers following use of alcohol hand rub.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqui Reilly, PhD, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Western Infirmary, Glasgow, United Kingdom

REFERENCES:
- [Derived] Reilly JS, Price L, Lang S, Robertson C, Cheater F, Skinner K, Chow A. A Pragmatic Randomized Controlled Trial of 6-Step vs 3-Step Hand Hygiene Technique in Acute Hospital Care in the United Kingdom. Infect Control Hosp Epidemiol. 2016 Jun;37(6):661-6. doi: 10.1017/ice.2016.51. Epub 2016 Apr 7. PMID 27050843